CLINICAL TRIAL: NCT03996031
Title: Plan to Thrive: Extending Cancer Survivorship Care Beyond the Clinic Using a Smartphone-enabled Monitoring, Navigation and Tailored Intervention Program
Brief Title: Plan to Thrive: Extending Cancer Survivorship Care Beyond the Clinic
Acronym: PTT
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Vignet, Inc. (Unknown)
Responsible Party: Principal Investigator, Sofia Garcia, Associate Professor, Northwestern University
Other Study IDs: STU00209558
Record Dates: First submitted 2019-06-19; First posted 2019-06-24 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Cancer, Breast; Cancer of Colon; Cancer of Rectum; Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Sample: All participants in this single-arm pilot study will receive access to Plan to Thrive. This mobile care management program is comprised of modules including educational interventions, health behavior trackers containing built-in reminders, symptom monitoring, and navigator services (see attached content). Access to intervention modules and individualized navigator services according to patients' needs as captured by 1) their patient-reported outcome (PRO) assessments via Plan to Thrive's symptom monitoring feature, and 2) patient requests. Following the baseline assessment, participants will engage with the Plan to Thrive app for a 90-day period.
  Interventions: Device: Plan to Thrive smartphone application

INTERVENTIONS:
Device: Plan to Thrive smartphone application — All participants in this single-arm pilot study will receive access to Plan to Thrive. This mobile care management program is comprised of modules including educational interventions, health behavior trackers containing built-in reminders, symptom monitoring, and navigator services (see attached content). Access to intervention modules and individualized navigator services according to patients' needs as captured by 1) their patient-reported outcome (PRO) assessments via Plan to Thrive's symptom monitoring feature, and 2) patient requests.

SUMMARY:
The purpose of this study is to test the usability of the Plan To Thrive smartphone application with cancer survivors. This study will involve three visits (baseline, follow-up, and feedback assessments). Between the baseline and follow-up time points, patients will undergo a 90-day period in which they will engage with app content. It is hypothesized that cancer survivors in this study will find the smartphone application, Plan to Thrive, an acceptable and feasible way to access post-treatment information. In addition, the investigators will explore preliminary efficacy by examining changes over time in primary (patient activation, patient knowledge and adherence to follow-up care recommendations and health behaviors) and secondary outcomes [symptom burden, health-related quality of life and patient satisfaction].

ELIGIBILITY:
INCLUSION CRITERIA:

* At least 18 years of age or older
* Prior history of cancer
* Completion of primary cancer treatment (i.e., surgery, chemotherapy and/or radiation; but can be receiving hormonal treatment)
* Have an e-mail account and reliable broadband access to the Internet
* Able to read, understand, and speak English sufficiently to understand study questionnaires and consent form

EXCLUSION CRITERIA:

* Has a medical condition with a life expectancy of fewer than 12 months
* Physical or cognitive disability that would prohibit them from participating in study procedures
* Having prior inpatient psychiatric treatment, or overt signs of, severe psychopathology (e.g., psychosis, substance dependence, suicidality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult survivors of cancer (e.g., breast, colorectal), who have completed their primary cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of enrollment | 4 months (baseline to follow-up)
  The investigators will explore the feasibility of the study procedures by examining rates of enrollment (defined as the percent of eligible individuals who consent to participate).
Rate of retention | 4 months (baseline to follow-up).
  The investigators will explore the feasibility of the study procedures by examining rates of retention (defined as percent of consented participants who complete follow-up measures).
Rate of app usage | 4 months (baseline to follow-up).
  The investigators will explore the feasibility of the study procedures by examining rates of usage (e.g., number of days participants access Plan to Thrive, percentage of prompts read).
Patient knowledge and adherence to follow-up care recommendations and health behaviors | 4 months (baseline to follow-up).
  This outcome will be assessed through a Health Behaviors Measure designed by Dr. Garcia for use in survivorship care planning (SCP) studies. This 14-item measure uses a 5-point Likert response scale. The content corresponds to SCP, NCCN and ACS recommendations for cancer survivorship. The investigators have slightly modified and shortened that measure for the present study to ensure it covers all the survivorship concerns addressed by Plan to Thrive. All patients will complete this measure at T1 and T2, and as part of the Survivor Symptom Update in Plan to Thrive.
Patient activation | 4 months (baseline to follow-up).
  Patient activation will be assessed using the "Patient Activation Measure" short form. The 13-item short form of the Patient Activation Measure is a reliable, validated (0-100 point) scale that assesses patient knowledge, skill and confidence for self-management. This will be administered at baseline (T1) and follow-up (T2).

SECONDARY OUTCOMES:
Symptom burden | 4 months (baseline to follow-up).
  Symptom burden will be assessed with computer adaptive tests (CATs) from the PROMIS measurement system. PROMIS is an NIH-sponsored system for measuring patient-reported health status, including physical, mental, and social well-being. Participants will complete the PROMIS Anxiety, Depression, Fatigue, and Pain Interference computer adaptive tests (CATs), which administer the minimum number of items necessary to accurately measure patient-reported outcomes while minimizing participant burden. These measures have all demonstrated reliability, precision, and construct validity based on their correlation with legacy instruments. All participants will complete these measures at T1 and T2. In addition, short forms of these PROMIS measures will be used, along with select items (physical activity, nutrition, alcohol use) as part of the Survivor Symptom Update in Plan to Thrive.
Health-related quality of life (HRQoL) | 4 months (baseline to follow-up).
  HRQoL will be measured with the FACT-G7, administered at baseline (T1) and follow-up (T2). The four-item needs assessment measure was used in prior studies and is based on questions used in a clinical initiative at the RHLCCC, which assess participants' supportive care needs. Items assess in what areas participants need support and service (e.g., coping, managing stress).
Patient satisfaction | 4 months (baseline to follow-up).
  Patient satisfaction will be assessed using the System Usability Scale (SUS), adminstered at follow-up (T2) only. The System Usability Scale (SUS) is a simple, ten-item scale giving a global view of subjective assessments of usability. This ten-item scale has selected statements that cover a variety of aspects of system usability, such as the need for support, training, and complexity, and thus have a high level of face validity for measuring usability of a system. SUS is a Likert scale, which is based on forced choice questions, where a statement is made and the respondent then indicates the degree of agreement or disagreement with the statement on a 5 point scale. SUS yields a single number representing a composite measure of the overall usability of the system being studied. SUS scores have a range of 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia F Garcia, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No